CLINICAL TRIAL: NCT05864742
Title: A Phase II Study of Genetically Risk-Stratified Combination of Venetoclax, Ibrutinib and Rituximab (With and Without Navitoclax) in Patients With Relapsed and Refractory Mantle Cell Lymphoma (AIM2)
Brief Title: Genetically Risk-Stratified Venetoclax, Ibrutinib, Rituximab (± Navitoclax) in Relapsed/Refractory Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/001
Record Dates: First submitted 2023-05-01; First posted 2023-05-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Mantle Cell Lymphoma Refractory
MeSH Terms: interventions — ibrutinib; venetoclax; navitoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-Risk Cohort (Experimental): Patients without the high-risk mutations (no 9p21.1-24.3 loss, no SMARCA2 or SMARCA4 mut/del) will be treated with ibrutinib, rituximab and venetoclax.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax; Drug: Rituximab
- High-Risk Cohort (Experimental): Patients with the high-risk mutations (9p21.1-24.3 loss, SMARCA2 and/or SMARCA4 mut/del) will be treated with ibrutinib, rituximab, venetoclax and navitoclax.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax; Drug: Navitoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — 560 mg daily continuously
  Other Names: imbruvica
Drug: Venetoclax — Oral daily. Dose escalation every 7 days (if no TLS) 20mg, 50mg, 100mg, 200mg and 400mg
  Other Names: Venclexta
Drug: Navitoclax — Oral daily. Dose-escalation every 14 days (if plt >75x10^9/L) 50mg, 100mg, 150mg, and 200mg (target dose)
  Other Names: ABT-263
  Arms: High-Risk Cohort
Drug: Rituximab — 375mg/m2, intravenous. To be given on day 1 of weeks 1, 2, 3, 4 of C1 and day 1 of C2-C8
  Other Names: Rituxan

SUMMARY:
This is an open label, multi-centre, phase II study in which RR MCL patients will be genetically risk-stratified into Standard risk (no 9p21.1-24.3 loss, no SMARCA2 or SMARCA4 mut/del) and High risk (9p21.1-24.3 loss, SMARCA2 and/or SMARCA4 mut/del).

Patients without the high-risk mutations will be treated with ibrutinib, rituximab and venetoclax. Patients with the high-risk mutations will be treated with ibrutinib, rituximab, venetoclax and navitoclax.

DETAILED DESCRIPTION:
The combination of ibrutinib and venetoclax in patients with RR MCL (50% TP53 aberrant) was explored in the AIM1 study. It demonstrated a CR rate of 71% (p<0.001) with an estimated 15 month PFS and 18-month OS of 78% and 74% respectively. Importantly, using ASO-PCR with sensitivity of 1 in 104-105, 56% of all patients and 82% of those who had achieved CR were MRD-negative. The combination was well tolerated with generally low-grade side effects including diarrhoea (83%), fatigue (75%) and nausea or vomiting (71%). Tumour lysis occurred in 8% (n=2) of the cohort. These results led to the initiation of a global phase III registration study comparing ibrutinib vs ibrutinib-venetoclax in patients with RR MCL (ClinicalTrials number NCT03112174).

The addition of anti-CD20 monoclonal antibodies (mAb) has significantly improved the outcomes in indolent and aggressive B-cell lymphomas. For instance, in Australia, the 5-year OS has improved from 53.4% in 1997 to 67.9% in 2007 largely due to incorporation of rituximab into the standard treatment regimens. In a phase II study of patients with RR MCL, the addition of rituximab to ibrutinib resulted in a considerably higher CR rate (44%) than with ibrutinib monotherapy (21%).The combination of an anti-CD20 mAb with a BTK and BCL-2 inhibitor was explored in the OSASIS study which combined obinutuzumab with ibrutinib and venetoclax in RR MCL (n=12). Venetoclax was administered at the dose range of 200-800mg.The combination resulted in high response rates and MRD-negativity in 77% of those who had achieved CR. Toxicities included haematological grade 3-4 AEs (58%), no dose limiting toxicity (DLT) and no clinically significant non-haematological Grade 3-4 AEs. However, it is unknown what the CR rate and MRD-negativity rates are in genetically defined risk groups in this small study.

Despite the encouraging results of AIM1, approximately 30% of patients failed to respond to the ibrutinib and venetoclax combination or relapsed whilst on study therapy after initially achieving CR. Genomic analysis of these patients in comparison to those who had sustained responses identified 9p21.1-24.3 loss or mutations in the SWI/SNF chromatin remodelling complex (SMARCA2 and/or SMARCA4 mut/del) as mechanisms of resistance through transcriptional upregulation of BCL-xL.20 This is a BCL2 family protein not targeted by venetoclax therefore providing a selective advantage against venetoclax-based therapy.

Navitoclax, a BCL2/BCL-XL/BCL-W inhibitor, was demonstrated by our in-vitro data to be able to overcome the resistance in SWI/SNF mutant cells, resensitising them to the ibrutinib-venetoclax combination.The combination of navitoclax and venetoclax has been recently explored in RR acute lymphoblastic leukaemia (ALL) and lymphoblastic lymphoma. Venetoclax was administered at 200mg on day 1 followed by 400mg daily thereafter. Navitoclax was administered at 3 dose levels (25mg, 50mg and if >45kg also 100mg). Common non-haematological AEs included diarrhoea (47%), nausea (47%), hypokalaemia (45%) and abdominal pain (43%) while Grade 3-4 haematologic AEs included febrile neutropenia (47%), thrombocytopenia (26%) and anaemia (17%). The incidence of grade 3-4 thrombocytopenia in this study is consistent with existing data on navitoclax toxicity profile. It is caused by navitoclax-mediated inhibition of Bcl-XL leading to accelerated platelet apoptosis. Combination with venetoclax allows for lower doses of navitoclax which can mitigate the effect on platelets.

Although there is no published data on the combination of navitoclax and rituximab, the safety and synergy of rituximab and navitoclax in CLL and indolent lymphoma has been reported with better response rates than in Phase I studies with either agent alone.

The AIM1 study demonstrated ibrutinib and venetoclax to be a highly effective treatment strategy for patients with RR MCL. Ancillary questions that we will address include:

1. Can addition of rituximab to the venetoclax and ibrutinib combination increase the depth and durability of response RR MCL?
2. Can addition of navitoclax in high-risk RR MCL improve rates of CR?
3. What is the safety and tolerability of these combinations?

The rationale for the staggered drug introduction and dose titration:

1. Ibrutinib and rituximab lead-in before venetoclax (and navitoclax in high-risk group):

   * Ibrutinib lead-in is expected to sensitise the lymphoma cells to venetoclax
   * Rituximab-induced rapid cytoreduction in order to reduce the tumour cell numbers and therefore the risk of patients harbouring MCL cells capable of adaption to the BH3-mimetics
   * Maintaining the same dosing schedule of ibrutinib and venetoclax as AIM1 in the standard-risk cohort would allow direct comparison with AIM1
2. Navitoclax dosing:

   * Given the ability of BCL-xL to be rapidly up-regulated in response to venetoclax and ibrutinib, co-administration of navitoclax and venetoclax is crucial. Navitoclax will therefore be introduced in week 4, i.e. after 3 weeks
   * We acknowledge that recovery of the platelet count whilst on navitoclax relies on compensatory mechanisms by the bone marrow, which may be suppressed by venetoclax, however, in order to effectively inhibit BCL-XL, we propose a target dose of 200mg with careful up-titration from an initial dose of 50mg as guided by the platelet count
   * Furthermore, recovery of navitoclax-induced thrombocytopenia would partially depend on the bone marrow reserve. Bone marrow involvement in MCL has been reported in 5029-63%30 of cases which is significantly lower than in CLL or ALL. We therefore anticipate that the impact of navitoclax on platelet count would be better compensated in MCL than in diseases with greater degree of bone marrow infiltration. Importantly, only 2 out of 24 patients (8%) on AIM1 study had a platelet count of <75 x 109/L at screening. Throughout the first 16 weeks, the platelet count remained >75 x 109/L in 92% and >50 x 109/L in 96% of patients (unpublished data)
   * Additionally, in order to mitigate the risk of ibrutinib-related bleeding exacerbated by Grade 3-4 thrombocytopenia, ibrutinib and navitoclax will be withheld until platelet count is ≥25 x 109/L and there is no further bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 years of age.
2. Patient must have a confirmed diagnosis of MCL according to World Health Organisation ([WHO] 2008) criteria, and have received at least one prior line of systemic therapy for their disease. Patients recently commenced on ibrutinib (≤4 weeks) will be allowed to enrol as long as at the time of enrolment there is measurable disease and no disease progression.
3. Patient requires treatment in the opinion of the investigator, and has at least one site of assessable disease not previously irradiated (such as lymph node with largest diameter ≥1.5cm, or unequivocal hepatomegaly/splenomegaly).
4. Patient has an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2 .
5. Patient must have adequate bone marrow function independent of growth factor support at screening as follows:

   * Absolute Neutrophil Count (ANC) ≥ 0.75 x 109/L (neutropenia due to marrow infiltration may be supported by growth factors)
   * Platelets ≥ 50 x 109/L (≥ 30 x 109/L if reduced counts due to marrow infiltration; entry platelet count must be independent of transfusion within 7 days)
6. Patients must have adequate coagulation, renal, and hepatic function, per laboratory reference range at screening as follows:

   * Activated partial thromboplastin time (aPTT) and prothrombin time (PT) ≤1.5 × the upper limit of normal (ULN)
   * Calculated creatinine clearance of at least 30 mL/min using the Cockcroft-Gault equation or a 24-hour urine collection (Appendix 2)
   * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤ 3.0 × ULN of institution's normal range
   * Bilirubin ≤1.5 × ULN. Patients with documented Gilbert's Syndrome may have a bilirubin > 1.5 × ULN
7. Female patients of childbearing potential and non-sterile male patients (with partner(s) of child bearing potential) must practice at least one of the following methods of birth control with partner(s) from initial study drug administration to 90 days after the last dose of study drug:

   * Total abstinence from sexual intercourse as the preferred life style of the patient; periodic abstinence is not acceptable
   * Surgically sterile partner(s); acceptable sterility surgeries are: vasectomy, bilateral tubal ligation, bilateral oophorectomy or hysterectomy
   * Intrauterine device
   * Double-barrier method (contraceptive sponge, diaphragm or cervical cap with spermicidal jellies or cream AND a condom)
   * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration
8. Female patients of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [B-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study.
9. Male patients must agree to refrain from sperm donation, from initial study drug administration until 90 days after the last dose of study drug.
10. Patient is able to swallow whole tablets.
11. Patient (or their legally acceptable representatives) must sign an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

1. Patient has undergone an allogeneic stem cell transplant within the last 6 months or currently has active graft-vs-host disease requiring the use of immunosuppressants.
2. Patient has active and uncontrolled autoimmune cytopenias (for 2 weeks), including autoimmune haemolytic anaemia and immune thrombocytopenic purpura.
3. Patient has current central nervous system (CNS) involvement by MCL.
4. Patient currently receiving ibrutinib for >4 weeks or previously received a Bruton's tyrosine kinase (BTK) inhibitor or B-cell lymphoma 2 (bcl-2) inhibitor.
5. Patient has received the following within 30 days prior to the first dose of study drug:

   • Monoclonal antibody given with anti-neoplastic intent
6. Patient has received any of the following within 14 days prior to the first dose of study drug, or has not recovered to less than CTCAE grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy:

   * Any anti-cancer therapy including chemotherapy, or radiotherapy
   * Investigational therapy, including targeted small molecule agents
7. Patient has received the following within 7 days prior to the first dose of study drug:

   • Steroid therapy given with anti-neoplastic intent
8. Patients requires ongoing therapy with:

   * Potent CYP3A inhibitors (such as indinavir, ketoconazole, and clarithromycin)
   * Potent CYP3A inducers (e.g., rifampin, phenytoin, carbamazepine or St. John's Wort)
   * Warfarin, or equivalent vitamin K antagonist
   * Antiretroviral medications.
9. Patient has consumed the following within 3 days prior to the first dose of study drug:

   * Grapefruit, or
   * Grapefruit products, or
   * Seville oranges (including marmalade containing Seville oranges), or
   * Star fruit
10. Patient has clinically significant cardiovascular disease such as uncontrolled arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
11. Patient has a life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of oral drugs, or put the study outcomes at undue risk:

    • Specifically, a patient with history of stroke or intracranial haemorrhage within 6 months prior to enrolment is excluded
12. Patient has a history of other active malignancies other than MCL within the past 2 years prior to study entry, with the exception of:

    * Adequately treated in situ carcinoma of the cervix uteri
    * Adequately treated basal cell carcinoma of the skin or localised squamous cell carcinoma of the skin
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
13. Patient has active Hepatitis C Virus (HCV) or active Hepatitis B Virus (HBV) infection or known history of human immunodeficiency virus (HIV) or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
14. Received live, attenuated vaccines within 4 weeks prior to the first dose of study drug.
15. Major surgery within 4 weeks prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Depth of MCL response to venetoclax and ibrutinib in combination with rituximab as determined by MRD at 16 weeks. | 2.5 years
  Standard risk MCL (no 9p21.1-24.3 loss, SMARCA2 or SMARCA4 mut/del): to evaluate the depth of response to venetoclax and ibrutinib in combination with rituximab in the treatment of patients with MCL, as determined by MRD clearance rate at 16 weeks.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peter MacCallum Cancer Centre, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No